CLINICAL TRIAL: NCT05978492
Title: A Multicenter, Open-label, Phase 1 Dose Escalation and Expansion Study of TXN10128, an Inhibitor of ENPP1 as Monotherapy and Combination Therapy With Irinotecan or Paclitaxel in Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of TXN10128 in Subjects With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Txinno Bioscience Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TXN10128-01
Record Dates: First submitted 2023-07-20; First posted 2023-08-07 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Locally Advanced (Unresectable) or Metastatic Solid Tumors
Keywords: ENPP1; ENPP1 inhibitor; TXN10128; TxinnoBio; Txinno Bioscience; Innate immune; STING pathway
MeSH Terms: interventions — Irinotecan; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Bayesian optimal interval (BOIN) design will be employed to find the MTD. The target DLT rate for determining the MTD is 30% for this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort A-1 (Experimental): TXN10128 Monotherapy Dose esclation part
  Interventions: Drug: TXN10128
- Cohort B-1 (Experimental): Combination Therapy with TXN10128 and Irinotecan Dose esclation part
  Interventions: Drug: TXN10128; Drug: Irinotecan
- Cohort C-1 (Experimental): Combination therapy with TXN10128 and Paclitaxel Dose esclation part
  Interventions: Drug: TXN10128; Drug: Paclitaxel

INTERVENTIONS:
Drug: TXN10128 — TXN10128: Oral administration once daily everyday
Drug: Irinotecan — Intravenous (IV) administration at 150 mg/m2 twice (Day 1 and Day 15) at intervals of 2 weeks in one cycle
  Arms: Cohort B-1
Drug: Paclitaxel — IV administration at 80 mg/m2 three times (Day 1, Day 8, and Day 15) at intervals of 1 week in one cycle (IV administration at 90 mg/m2 for patients with breast cancer)
  Arms: Cohort C-1

SUMMARY:
This is a phase I clinical trial to primarily evaluate the safety, tolerability, and addtionally assess pharmacokinetics, pharmacodynamics, and antitumor activity of investigational product, TXN10128. The target subjects will be consisted of patients with locally advanced (unresectable) or metastatic soild tumors.

This study includes a dose-escalation part and a dose-expansion part, and a TXN10128 monotherapy part and a TXN10128 + Irinotecan or Paclitaxel combination therapy part.

DETAILED DESCRIPTION:
This study includes a dose-escalation part and a dose-expansion part, and a TXN10128 monotherapy part and a TXN10128 + Irinotecan or Paclitaxel combination therapy part. The study includes dose-escalation and dose-expansion parts across three cohorts: TXN10128 monotherapy (Cohorts A) TXN10128 + Irinotecan (Cohorts B) and TXN10128+ Paclitaxel (Cohorts C).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥19 years of age at the time of informed consent.
* Histologically and/or cytologically confirmed any progressive, locally advanced (unresectable), or metastatic solid tumors that have relapsed or are refractory following the last line of treatment and for which prior standard therapy has been ineffective, or standard therapy does not exist or is not considered appropriate.
* ECOG performance status of 0 or 1.
* Life expectancy of at least 12 weeks.

Exclusion Criteria:

* Has leptomeningeal disease.
* Experienced a Grade ≥3 immune-related adverse events (irAE) with prior immunotherapy with the exception of non-clinically significant laboratory abnormalities.
* Prior organ transplantation.
* Known positive human immunodeficiency virus (HIV) infection.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
DLT | Day 1 up to Day 21 for Cohort A(TXN10128 mono cohort) and Day 1 up to Day 28 for Cohort B,C(TXN10128 combination with Irinotecan or paclitaxel cohort) in dose escalation period
  A DLT is defined as any of the following AEs (graded using NCI CTCAE v5.0) whose relationship to TXN10128 cannot be ruled out.
Adverse events (AE) | Up to 30 days from end of treatment
  Adverse events (AE) defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) criteria version 5.0 at each dose level

SECONDARY OUTCOMES:
Cmax | Up to 21 days from Day 1 dose
  The time to reach the maximum observed concentration (time)
AUC inf | Up to 21 days from Day 1 dose
  The area under the concentration-time curve extrapolated to infinity (mass*time/volume)
AUC last | Up to 21 days from Day 1 dose
  The area under the concentration (AUC) -time curve calculated to the last quantifiable concentration point (mass* time/volume)
Tmax | Up to 21 days from Day 1 dose
  The time to reach the maximum observed concentration (time)
T1/2 | Up to 21 days from Day 1 dose
  Elimination half-life, determined as 0.693/Lambda_z (time)
Vss | Up to 21 days from Day 1 dose
  Volume of distribution during the steady state phase (volume)
Best overall response (BOR) | Up to 30 days from end of treatment
  Best overall response will be summarized
Progression free survival (PFS) | Up to 30 days from end of treatment
  The survival function will be estimated using the Kaplan-Meier product limit method. Median duration, with a two-sided Brookmeyer-Crowley 90% confidence interval and Kaplan-Meier estimates of survival proportions will be provided at specified time points.
Disease control rate (DCR) | Up to 30 days from end of treatment
  The disease control rate is calculated as the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease
Duration of Response (DOR) | Up to 30 days from end of treatment
  Duration of response is defined as the time from the date of the first documented response (CR or PR), to the date of first documented progression, or death due to study indication. Estimates will use Kaplan-Meier method
Overall response rate (ORR) | Up to 30 days from end of treatment
  Overall response rate will be summarized with accompanying 90% exact binomial confidence interval (CI).

CONTACTS AND LOCATIONS:
Overall Officials: Min-Hee Ryu, M.D., Ph.D., Principal Investigator — Asan Medical Center; Do-Youn Oh, M.D., Ph.D., Principal Investigator — Seoul National University Hospital; Jin Seok Ahn, M.D., Ph.D., Principal Investigator — Samsung Medical Center; SeHyun Kim, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital; Ki-hyeong Lee, M.D., Ph.D., Principal Investigator — Chungbuk National University Hospital; Joo-Hwan Park, M.D., Ph.D., Principal Investigator — eoul National University Hospital
Locations (6):
- South Korea (6):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chungbuk National University Hospital, Cheonju, North Chungcheong
  - Seoul National Univ. Hospital, Seoul, Seoul
  - Asan Medical Center, Seoul, Seoul
  - Gachon University Gil Medical Center, Incheon
  - SAMSUNG Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Homepage of Txinno Bioscience — http://www.txinno.com